CLINICAL TRIAL: NCT07164274
Title: Prevalence of Gastroesophageal Reflux Disease, Its Association With Eating Behavior and Psychological Disturbance, and Its Impact On Quality Of Life, Among Medical Students In The MENA Region, A Multinational Cross-Sectional Study
Brief Title: Prevalence of GERD, Its Effect on HRQL and Psychological Disturbance, and the Effect of Eating Behaviors on GERD Prevalence
Status: Active, not recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Abdelmonam Mamdouh Abdelmonam Mohamed Ahmed Hagag, Dr, Zagazig University
Other Study IDs: ZU-IRB# 1580/5-Aug-2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gastro -Oesophagal Reflux; Eating Behavior Disorders
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: Questionnaire — An online questionnaire that will be shared via online platforms for medical students and interns in the Middle East countries to fill.

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common gastrointestinal disease. It is a chronic condition that is characterized by the regurgitation of stomach contents into the esophagus and is associated with heartburn. The occurrence of these symptoms for at least two weeks increases the likelihood of having GERD. Other GERD symptoms include chest pain, nausea, dysphagia, burping, water brash, and vomiting. All these symptoms negatively affect the patients' quality of life. The pathophysiology of GERD is multifactorial. Several factors have been suggested to cause GERD, including a hypotensive lower esophageal sphincter (LOS) and a defect in the gastric sling/clasp muscle fiber component.

The global prevalence of GERD is about 13.98% with variation among different countries and ethnic groups. In East Asia, it ranges from 2.5% to 7.5%, 8.5 to 25.9% in Europe, 18.1% to 27.8% in South and North America, and about 11.6% in Australia. In the Middle East, it ranges from 8.7% to 33.1%.

Several risk factors have been identified that increase the likelihood of having GERD. Obesity was found to be one of the risk factors that increases GERD. Also, dietary habits such as spicy food, coffee drinks, or administering NSAIDs increase the prevalence of having GERD.

On the other hand, psychological factors also play an important role in GERD severity. Both stress and anxiety are linked to an increase in GERD. A previous study showed that stress can increase heartburn symptoms in patients with heartburn and also increase in anxiety level was associated with an increase in esophageal reflux. Finally, depression was found to be associated with GERD, which can be explained by a change in the eating behavior in depressed patients.

Rationale Medical students suffer from a study burden, which increases their level of anxiety and stress. They also have a higher likelihood of having trouble with eating behavior or having a lot of coffee daily. This increases their likelihood of having GERD. In the Middle East, fewer studies have assessed the effect of GERD. A recent cross-sectional study assessed the prevalence of GERD among medical students in Egypt. They found a prevalence of 17.1%. They found an association between increasing stress levels and increasing GERD severity. Also, smoking was a significant risk factor for GERD symptoms. Another cross-sectional study among medical students in 21 universities in Egypt. They reported a prevalence of 28.4%. Again, they found that an increasing level of stress and anxiety was associated with increasing GERD severity. Finally, Two cross-sectional studies were conducted in Saudi Arabia. They reported a prevalence of 23.8% and 23.1% respectively. To our knowledge, no study has assessed the GERD and its related quality of life among medical students in Middle East and linked their findings with eating behaviour

ELIGIBILITY:
Inclusion Criteria:

* Medical students and interns studying medicine in the Middle East countries
* Have access to online platforms

Exclusion Criteria:

* Students or interns who refused to participate

Ages: 18 Years to 27 Years | Sex: All
Age Groups: Adult
Study Population: Medical students and interns in the Middle East countries
Sampling Method: Non-Probability Sample
Enrollment: 3773 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
GERD prevalence | through study completion, an average of 6 months
  The GERDQ questionnaire will be used. It is composed of 6 Likert scale questions that ask about GERD symptoms such as heartburn, nausea, and regurgitation. Each question has 4 answers scored from 0 to 3, making a rank from 0 to 18. If the participant scores 8 or more, this diagnosis is GERD. Furthermore, the severity can be assessed. A score of 0-2 makes 0 % of having GERD, 3-7 makes a 50% likelihood of having GERD, 8-10 makes a 79% and 11-18 makes a 89% of having GERD. This questionnaire has a sensitivity being 65% and a specificity being 71% to diagnose GERD
GERD_HRQL | through study completion, an average of 6 months
  The GERD-HRQL was used. This is a 16 Likert scale questionnaire that asks about the effect of GERD symptoms on the quality of life. The first 15 questions had 6 answers, ranging from no symptoms to Symptoms that are incapacitating - unable to do daily activities. This score ranges from 0 to 5. The sixteenth question asks about the present condition. The quality of life is calculated via the first 15 questions (scores from 0 to 75), with higher scores indicating lower quality of life.

SECONDARY OUTCOMES:
Eating behavior disorder | through study completion, an average of 6 months
  The Dutch Eating Behavior Questionnaire (DEBQ) was used. This is a 33 Likert scale questionnaire that assesses the eating behavior in three items (retained eating, emotional eating, and External eating). Each question is composed of 5 answers (from never to very often) and scores range from 1 to 5
Psychological disturbance | through study completion, an average of 6 months
  the DASS-21 was uses questionnaire. This is composed of 21 Likert scale questions, each had 4 answers scored from 0 to 3. The scale is divided into 3 sections to assess depression, stress, and anxiety. The cumulative score for each part will be multiplied by two for interpretation of the severity of each section.
  1. For the Depression score, 0-9 indicates a normal person, 10-13 indicates mild symptoms, 14-20 indicates moderate, 21-27 indicates severe symptoms, and 28+ indicates extremely severe symptoms.
  2. For anxiety scores, 0-7 indicates a normal person, and (8-9), (10-14), (15-19), and 20+ indicate mild, moderate, severe, and extremely severe levels of anxiety.
  3. For stress scores, 0-14 indicates a normal person. A score of (15-18), (19-25), 26-33), and 34+ indicate a mild, moderate, severe, and extremely severe levels of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of Medicine and Affiliated Hospital, Zagazig, Egypt

REFERENCES:
- [Result] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT07164274/Prot_SAP_000.pdf